CLINICAL TRIAL: NCT02164682
Title: The Effect of Caudal Block on the Postoperative Complications in Pediatric Patients After Hypospadias Repair
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0294
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Hypospadias
Keywords: Hypospadias repair; Caudal block; Postoperative complications
MeSH Terms: conditions — Hypospadias; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IV PCA group
  Interventions: Procedure: IV PCA group
- IV PCA+ caudal block group
  Interventions: Procedure: IV PCA+ caudal block group

INTERVENTIONS:
Procedure: IV PCA group — The IV PCA is performed by injecting fentanyl 15 mcg/kg with the following regimen
  Groups: IV PCA group
Procedure: IV PCA+ caudal block group — The IV PCA is performed by injecting fentanyl 15 mcg/kg with the following regimen + caudal block was 0.15% ropivacaine 1.2 cc/kg; a total volume of 100 cc, basal 2 cc, bolus 0.5 cc, and lockout time 15 minutes.)
  Groups: IV PCA+ caudal block group

SUMMARY:
Hypospadias refers to a disease represented by a congenital defect in the urethra meatus (urinary opening) in male children. Due to the postoperative pain, symptoms such as discomfort, agitation, and restlessness are generally found. In particular, young children with restlessness often express their pain or discomfort with their bodies because they are unable to express it in words. This severe restlessness may make an operated region unstable, accompanying bleeding, infection, or other surgery-related complications. Because postoperative pain control is very important, neuraxial block techniques such as epidural block or caudal block have been employed in addition to a penile dorsal nerve block. Although the neuraxial block technique including the caudal block is an easy and safe method and has an excellent effect, the neuraxial block technique poses a potential risk in the procedure. In addition, with respect to the surgical prognosis, it has been reported that penile engorgement may cause penile vasodilation, resulting in oozing at the surgical region or other surgical complications. However, there has not been a report on the increase of postoperative complications by penile vasodilation or on the difference in the recovery or surgical prognosis according to the types of pain control for young patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who underwent the tubularized incised plate (TIP) repair under hypospadias at our institution between January, 2010 and December, 2014

Exclusion Criteria:

* Patients whose medical records could not be analyzed for having undergone the first hypospadias surgery at another institution. Other exclusion criteria were as follows: over the age of 8 years, planned two-stage hypospadias repair, receiving continuous epidural analgesia, and without hypospadias as the final diagnosis.

Max Age: 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients who underwent the first hypospadias surgery at our institution between January, 2010 and December, 2014 (for 5 years).
Sampling Method: Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The postoperative complications related hypospadias repair | within 6 months after hypospadias repair
  The electronic medical records of pediatric patients who underwent hypospadias repair will be reviewed to analyze the difference in postoperative complications within 6 months after surgery between patients whose postoperative pain control was performed only by IV PCA and patients whose postoperative pain control was performed by caudal block combined with IV PCA.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University Health System, Seoul, Seoul, South Korea